CLINICAL TRIAL: NCT02241317
Title: Effects of Training of Medical Staff on the Outcome of In-Patients With Diabetes Mellitus on Regular Wards
Brief Title: Diabetes Mellitus at the University Medical Center of Mannheim
Acronym: DmUMM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Alexander Lammert, Dr. med. Alexander Lammert, Universitätsmedizin Mannheim
Other Study IDs: 2014-831R-MA
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus; Hypoglycaemia
Keywords: Diabetes mellitus; Hypoglycaemia; staff training; Education; blood glucose
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Development of a training concept for health care professionals (nursing and medical staff), according to the current guidelines on treatment of in-patients with Diabetes. Primary endpoint is the change in hypoglycaemia rates comparing data before and after the training. Hereby we can derive the effects of staff training on the quality of health care in this patient population.

DETAILED DESCRIPTION:
The prevalence of Diabetes in in-patients is about 32% and therefore exceeds significantly the prevalence in general population.

In most cases Diabetes is only a secondary diagnosis the medical staff has to deal with daily. The diagnosis which leads to hospital admission and the often multiple comorbidities complicate the metabolic control. Blood sugar imbalances present an additional risk for these patients and increase in-hospital mortality, length of hospital stay and general complications as nosocomial infections.

To improve hospital care for diabetics the Endocrine Society and the American College of Physicians published new guidelines on blood glucose management for non-ICU wards. Primarily they contain recommendations for blood glucose target range and standards to improve inpatient hospital care like standard operating procedures for blood glucose monitoring as well as hyper- and hypoglycaemic disturbances through to discharge management.

We developed a training concept for health care professionals (nursing and medical staff), according to the current guidelines on treatment of in-patients with Diabetes. Primary endpoint is the change in hypoglycaemia rates comparing data before and after the training. Hereby we can derive the effects of staff training on the quality of health care in this patient population.

So far there was only one comparable study published which showed a significant improvement of treatment quality by reducing hypoglycaemia rates considerably . The results of this study cannot be transferred due to substantial structural differences. More over there are no national diabetes management guidelines for inpatient treatment in Germany.

The following data will be collected:

* Anthropometric data (Age, Sex, Bodyweight, Height)
* Diagnosis
* POCT blood glucose values
* Other laboratory values
* Length of hospital stay

This study conforms to the requirements of the Declaration of Helsinki, Revision of 1996.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-Patients with Diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Hypoglycaemia | 2013-2015 (two years)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lammert, Dr. med., Principal Investigator — Universitätsmedizin Mannheim